CLINICAL TRIAL: NCT05548062
Title: Prospective Observational Study to Identify and Describe Predictive Factors for Thromboembolic Events in Patients With High-risk Polycythemia Vera
Brief Title: Study to Identify and Describe Predictive Factors for Thromboembolic Events in Patients With High-risk Polycythemia Vera
Acronym: Prospero
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424BIT01
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Polycythemia Vera
Keywords: polycythemia vera; high-risk polycythemia vera; PV; Ruxolitinib; NIS; Italy; TE; predictive factors; hydroxyurea
MeSH Terms: conditions — Polycythemia Vera | interventions — Hydroxyurea; ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hydroxyurea: Patients being treated with hydroxyurea at enrollment and for at least 18 months prior to enrollment. Patients may switch to ruxolitinib treatment during the study in case of inadequate response or intolerance.
  Interventions: Other: Hydroxyurea
- Ruxolitinib: Patients on treatment with ruxolitinib who started treatment up to 18 months prior to enrollment.
  Interventions: Other: Ruxolitinib

INTERVENTIONS:
Other: Hydroxyurea — Prospective observational study. There is no treatment allocation. Patients prescribed with Hydroxyurea are eligible to enroll into this study.
  Groups: Hydroxyurea
Other: Ruxolitinib — Prospective observational study. There is no treatment allocation. Patients prescribed with Ruxolitinib are eligible to enroll into this study.
  Groups: Ruxolitinib

SUMMARY:
This is a prospective observational study that will enroll patients with high-risk Polycythemia Vera (PV) with at least one Thromboembolic Event (TE) after diagnosis or up to 2 years prior to diagnosis.

This is a non-randomized study, and to ensure a sufficient number of patients in both cohorts, enrollment in each cohort will be terminated once the target of 150 patients has been reached.

DETAILED DESCRIPTION:
All patients are already on treatment with hydroxyurea or ruxolitinib at enrollment as per clinical practice and independently of their participation in this study. In addition, the follow-up visits and the evaluation procedures required in the study protocol correspond to current clinical practice. According to local regulations related to observational studies, assessments such as blood tests are justified by the purpose and rationale of the study (i.e., the identification of possible predictive factors of TEs) and are considered current clinical practice. Data related to other procedures will be collected only if such procedures are performed as per clinical practice but are not required otherwise.

Patients in both cohorts will be followed for 3 years after enrollment and will have visits at Months 6, 12, 18, 24, 30 and 36. A time window of ± 1 month is permitted for all visits.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Age ≥18 years.
3. Diagnosis of PV according to WHO 2008 or WHO 2016 and high-risk stratification according to European LeukemiaNet (ELN) classification.
4. At least one TE after diagnosis or up to 2 years prior to diagnosis.
5. Patients on treatment with hydroxyurea at enrollment and for at least 18 months prior to enrollment or those on treatment with ruxolitinib who started treatment up to 18 months before enrollment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve patients in Italy with high-risk Polycythemia Vera
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of abnormalities presented in patients with Thromboembolic Events (TEs) during the follow up | Up to 36 months
  Demographics, blood pressure, laboratory blood tests, and use of antiplatelets and/or anticoagulants are predictors of TE occurrence, a univariate Cox regression model for repeated events will be applied for each predictor considering all the TEs occurring within 12 months and the time from baseline to each occurrence. Predictors found statistically significant at the 5% level will then be considered in a multivariate Cox regression model for repeated events.
Blood pressure | Up to month 36
  Blood pressure is going to be collected
Number of patients with abnormal Body Mass Index (BMI) | Up to month 36
  Number of patients with abnormal Body Mass Index (BMI) will be collected
Number of patients with abnormal weight | Up to month 36
  Number of patients with abnormal weight will be collected
Number of patients with abnormal Neutrophil (NEP) count | Up to 36 months
  Number of patients with abnormal Neutrophil (NEP) count will be collected
Number of patients with abnormal White blood Count (WBC) | Up to 36 months
  Number of patients with abnormal White blood Count (WBC) will be collected
Number of patients with abnormal Lymphocytes (LYP) count | Up to 36 months
  Number of patients with abnormal Lymphocytes (LYP) count will be collected
Number of participants using antiplatelets and/or anticoagulants on the incidence of TEs | Up to 36 months
  Number of participants using antiplatelets and/or anticoagulants on the incidence of Thromboembolic Events (TEs) will be collected

SECONDARY OUTCOMES:
Synergistic combinations of predictive factors | Up to 36 months
  Synergistic combinations of predictive factors (Red cell Distribution Width, neutrophils, lymphocytes, neutrophil/ lymphocyte ratio and platelets).
  Synergy score is defined as the product of the individual significances of variable 1 and 2 (expected) divided by the significance of the two-variable model (observed) To investigate cases of extreme synergy, instances in which two variables split the given cohort into high-risk and low-risk patients are far better than either variable alone. A simple synergy scoring metric to rank variable in terms of synergy (S):S12=(P1*P2)/P12 where P1 and P2 are the maximum possible (Cox regression derived) p-values for variable 1 and variable 2 and P12 was the max. p-value possible from the combination of variables 1 and 1. This synergy is intended to capture a variable that may provide exclusive non-redundant information when attempting to split a cohort based on risk and may provide an added insight into the functional/clinical rationale of a model
Yearly incidence of TEs | 36 months
  Yearly incidence of Thromboembolic Events (TEs) will be collected
Incidence of arterial and venous TEs in the hydroxyurea and ruxolitinib cohorts | 36 months
  Incidence of arterial and venous TEs in the hydroxyurea and ruxolitinib cohorts will be collected
Incidence and severity of adverse events | 36 months
  Incidence and severity of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- Italy (30):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Como, CO
  - Novartis Investigative Site, Cosenza, CS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Tricase, LE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Pagani, SA
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Viterbo, VT
  - Novartis Investigative Site, Napoli

IPD SHARING:
Plan to Share IPD: No